CLINICAL TRIAL: NCT00368251
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel Study to Evaluate the Efficacy and Safety of Brivaracetam Used as Adjunctive Treatment for 12 Weeks in Adolescent and Adult Patients (≥ 16 Years) With Genetically Ascertained Unverricht-Lundborg Disease
Brief Title: Brivaracetam as add-on Treatment of Unverricht-Lundborg Disease (ULD) in Adolescents and Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: N01236; 2006-001536-46 (EudraCT Number)
Expanded Access: NCT03532516 (Available)
Record Dates: First submitted 2006-08-23; First posted 2006-08-24 (Estimated); Results first posted 2016-04-13 (Estimated); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Unverricht-Lundborg Disease
Keywords: Unverricht-Lundborg Disease; Baltic Myoclonus; Progressive Myoclonic Epilepsies; Myoclonus; Brivaracetam
MeSH Terms: conditions — Unverricht-Lundborg Syndrome; Myoclonic Epilepsies, Progressive; Myoclonus | interventions — brivaracetam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo Placebo twice a day (bid), 14 weeks (2 week Up-Titration Period + 12 week Maintenance Period)
  Interventions: Other: Placebo
- Brivaracetam 5 mg/day (Experimental): Brivaracetam (BRV) 5 mg/day 5 mg twice a day (bid) using 2.5 mg tablets for 12 weeks (after 2 week Up- Titration Period)
  Interventions: Drug: BRV 2.5 mg
- Brivaracetam 150 mg/day (Experimental): Brivaracetam (BRV) 150 mg/day 150 mg twice a day (bid) using 25 mg and 50 mg tablets for 12 weeks (after 2 week Up-Titration Period)
  Interventions: Drug: BRV 25 mg; Drug: BRV 50 mg

INTERVENTIONS:
Other: Placebo — * Pharmaceutical Form: Tablet
  * Concentration: 2.5 mg, 25 mg and 50 mg
  * Route of Administration: Oral use
  Arms: Placebo
Drug: BRV 2.5 mg — * Pharmaceutical Form: Tablet
  * Concentration: 2.5 mg
  * Route of Administration: Oral use
  Other Names: ucb34714
  Arms: Brivaracetam 5 mg/day
Drug: BRV 25 mg — * Pharmaceutical Form: Tablet
  * Concentration: 25 mg
  * Route of Administration: Oral use
  Arms: Brivaracetam 150 mg/day
Drug: BRV 50 mg — * Pharmaceutical Form: Tablet
  * Concentration: 50 mg
  * Route of Administration: Oral use
  Arms: Brivaracetam 150 mg/day

SUMMARY:
The study will compare the efficacy and safety of Brivaracetam with placebo in patients with Unverricht- Lundborg Disease (ULD).

ELIGIBILITY:
Inclusion Criteria:

- Subjects with diagnosed Unverricht-Lundborg disease (ULD) ascertained by appropriate genetic testing for a homozygous or compound heterozygous mutation in the CSTB gene- Subjects with moderate to severe myoclonus documented by an Action Myoclonussum score of ≥ 30 (evaluation by investigator)-Subjects currently being or having been treated with clonazepam up to the maximum recommended daily dose of 20 mg or up to their individual optimal dose as assessed by the investigator- Subjects currently being or having been treated with valproate up to the maximum recommended daily dose 60 mg/kg or serum levels of 100 mcg/ml or up to their individual optimal dose as specified by the investigator- Male/female subjects from 16 years onwards. Subjects under 18 years may only be included where legally permitted and ethically accepted

Exclusion Criteria:

- Subjects currently on felbamate or having been on felbamate within less than 18 months prior to Visit 1- Subjects currently treated with phenytoin or having been on phenytoin in the last month prior to Visit 1- Subjects currently on vigabatrine. Subjects having been on vigabatrine if no visual fields examination report available including standard static (Humphrey or Octopus) or cinetic perimetry (Goldman)- Subject taking any drug with possible central nervous system (CNS) effects- Subjects taking any drug that may significantly influence the metabolism of BRV (CYP2C or CYP3A potent inducers/inhibitors)- Known clinically significant acute or chronic illness or illness which may impair reliable participation in the trial, necessitate the use of medication not allowed by protocol or represent a safety risk in the Investigator's opinion- Subjects with history of severe adverse hematological reaction to any drug- Impaired hepatic function: ALAT/SGPT, ASAT/SGOT, alkaline phosphatase, GGT value of more than three times the upper limit of the reference range- History of suicide attempt during the last 5 years- Subject with suicidal ideations within the last year or at risk of suicide attempt unless cleared by written confirmation from a psychiatrist and approved by the UCB physician- Ongoing psychiatric disorder other than mild controlled disorder

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2006-11; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (18):
- United States (4):
  - 135, San Francisco, California
  - 133, Gainesville, Florida
  - 132, New York, New York
  - 131, Charlottesville, Virginia
- Canada (3):
  - 151, Vancouver, British Columbia
  - 150, Montreal, Quebec
  - 152, Québec, Quebec
- 100, Helsinki, Finland
- France (3):
  - 122, Bron
  - 121, Lille
  - 120, Paris
- 170, Tel Aviv, Israel
- Russia (3):
  - 141, Moscow
  - 142, Saint Petersburg
  - 143, Samara
- Serbia (2):
  - 161, Belgrade
  - 162, Belgrade
- 180, Manouba, Tunisia

REFERENCES:
- [Derived] Ben-Menachem E, Baulac M, Hong SB, Cleveland JM, Reichel C, Schulz AL, Wagener G, Brandt C. Safety, tolerability, and efficacy of brivaracetam as adjunctive therapy in patients with focal seizures, generalized onset seizures, or Unverricht-Lundborg disease: An open-label, long-term follow-up trial. Epilepsy Res. 2021 Feb;170:106526. doi: 10.1016/j.eplepsyres.2020.106526. Epub 2020 Dec 4. PMID 33461041
- [Derived] Kalviainen R, Genton P, Andermann E, Andermann F, Magaudda A, Frucht SJ, Schlit AF, Gerard D, de la Loge C, von Rosenstiel P. Brivaracetam in Unverricht-Lundborg disease (EPM1): Results from two randomized, double-blind, placebo-controlled studies. Epilepsia. 2016 Feb;57(2):210-21. doi: 10.1111/epi.13275. Epub 2015 Dec 15. PMID 26666500
- See also: Product Information — https://www.briviact.com/briviact-PI.pdf?v=1479491757
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 72 subjects were screened, 56 subjects were randomized. Participant Flow refers to all subjects randomized who are identical with the Intent-To-Treat (ITT) Population, which consists of all randomized subjects who took at least one dose of study medication.
Groups:
- Placebo: Placebo twice a day (bid), 14 weeks (2 week Up-Titration Period + 12 week Maintenance Period)
- Brivaracetam 5 mg/Day: Brivaracetam (BRV) 5 mg/day 2.5 mg twice a day (bid) using 2.5 mg tablets for 12 weeks (after 2 week Up- Titration Period)
- Brivaracetam 150 mg/Day: Brivaracetam (BRV) 150 mg/day 75 mg twice a day (bid) using 25 mg and 50 mg tablets for 12 weeks (after 2 week Up-Titration Period)
Period: Overall Study
Arm/Group | Placebo | Brivaracetam 5 mg/Day | Brivaracetam 150 mg/Day
Started | 18 | 20 | 18
Completed | 17 | 20 | 17
Not Completed | 1 | 0 | 1
Not completed — SAE, non-fatal | 1 | 0 | 0
Not completed — AE, non-serious non-fatal | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Baseline Analysis Population contains all randomized subjects who are identical with the Intent-To-Treat (ITT) population.
Arm/Group | Placebo | Brivaracetam 5 mg/Day | Brivaracetam 150 mg/Day | Total Title
Number analyzed (Participants) | 18 | 20 | 18 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1 | 2
  Between 18 and 65 years | 18 | 19 | 17 | 54
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.3 (9.2) | 35.8 (10.9) | 33.7 (11.4) | 34.65 (10.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 9 | 32
  Male | 6 | 9 | 9 | 24
Region of Enrollment [Number; unit: participants]
  Serbia | 2 | 2 | 2 | 6
  France | 3 | 2 | 3 | 8
  United States | 2 | 3 | 4 | 9
  Canada | 4 | 3 | 2 | 9
  Finland | 3 | 4 | 2 | 9
  Russian Federation | 2 | 3 | 3 | 8
  Israel | 0 | 0 | 2 | 2
  Tunisia | 2 | 3 | 0 | 5

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline to the End of Treatment Period on the Action Myoclonus Score (Unified Myoclonus Rating Scale (UMRS) Section 4)
Description: The range for Action Myoclonus Score (centrally read) is 0 (best) - 160 (worst). Percent change from Baseline = 100 X ((Baseline UMRS4 - Treatment UMRS4) / Baseline UMRS4). Baseline is defined as the last non-missing value prior to or on Randomization Visit.
Time Frame: From Baseline to End of Treatment Period (Week 14 or Early Discontinuation Visit)
Population: The number of subjects is equal to the number of subjects in the Intent-To-Treat (ITT) population having non-missing post-baseline results for the percent change from baseline on the functional disability score (UMRS section 5). In case a subject drops out, the result at Early Discontinuation Visit is used.
Measure: Median (Full Range); unit: Percent change
Arm/Group | Placebo | Brivaracetam 5 mg/Day | Brivaracetam 150 mg/Day
Number analyzed (Participants) | 18 | 20 | 18
Percent change | 17.45 [-170.0 to 61.5] | -4.60 [-430.0 to 81.8] | 12.34 [-58.3 to 96.9]
Statistical Analysis 1: Comparison: Placebo vs Brivaracetam 150 mg/Day; The first hypothesis for the primary efficacy variable compares placebo versus Brivaracetam (BRV) 150 mg/day. The second hypothesis for the primary efficacy variable compares placebo versus BRV 5 mg/day. However, this second hypothesis will only be tested when all the hypotheses for placebo versus BRV 150 mg/day are significant for the primary three UMRS related secondary endpoints. The hypotheses will be tested using nonparametric analysis. The study was designed to have 80 % power; Test type: Superiority or Other; p = 0.942, stratified Wilcoxon Test — All hypotheses are tested at the 5 % level. The multiplicity scheme (hierarchical testing procedure) assures strong control of the type I error at the 5 % level; Estimates and confidence intervals from Hodges-Lehmann (unstratified); Hodges-Lehmann-estimator of difference = 0.15, 95% CI 2-sided [-26.12 to 24.96] — Difference versus Placebo was calculated
Statistical Analysis 2: Comparison: Placebo vs Brivaracetam 5 mg/Day; Test type: Superiority or Other; p = 0.105, stratified Wilcoxon Test — Tested at the 5 % level - given the primary endpoint and the three UMRS related secondary endpoints comparing placebo versus Brivaracetam (BRV) 150 mg/day are significant at the 5 % level (hierarchical testing procedure); Estimates and confidence intervals from Hodges-Lehmann (unstratified); Hodges-Lehmann-estimator of difference = -18.05, 95% CI 2-sided [-39.31 to 4.86] — Difference versus Placebo

2. Secondary Outcome: Percent Change From Baseline to the End of Treatment Period on the Functional Disability Score (Unified Myoclonus Rating Scale (UMRS) Section 5)
Description: The range for Functional Disability Score is 0 (best) to 28 (worst). Percent change from Baseline = 100 X ((Baseline UMRS5 - Treatment UMRS5) / Baseline UMRS5). Baseline is defined as the last non-missing value prior to or on Randomization Visit.
Time Frame: Baseline to End of Treatment Period (Week 14 or Early Discontinuation Visit)
Population: as for outcome 1
Measure: Median (Full Range); unit: Percent change
Arm/Group | Placebo | Brivaracetam 5 mg/Day | Brivaracetam 150 mg/Day
Number analyzed (Participants) | 18 | 20 | 18
Percent change | 0.00 [-380.0 to 53.8] | 0.00 [-380.0 to 60.0] | 0.00 [-85.7 to 75.0]
Statistical Analysis 1: Comparison: Placebo vs Brivaracetam 150 mg/Day; If primary efficacy is proven for Brivaracetam (BRV) 150 mg/day, the following secondary endpoints will be tested for Placebo versus BRV 150 mg/day. The testing scheme will be hierarchical, thus statistical significance at 5 % on BRV 150 mg/day on a secondary endpoint is needed to continue testing BRV 150 mg/day at 5 % significance level for the next secondary endpoint; Test type: Superiority or Other; p = 0.672, stratified Wilcoxon Test — Tested at the 5 % level - given the Primary Outcome testing Placebo versus BRV 150 mg/day is significant at the 5 % level (hierarchical testing procedure); Estimates and confidence intervals are obtained from Hodges-Lehmann(unstratified); Hodges-Lehmann-estimator of difference = 1.24, 95% CI 2-sided [-21.90 to 31.06] — Difference versus Placebo
Statistical Analysis 2: Comparison: Placebo vs Brivaracetam 5 mg/Day; In case the three endpoints are significant for placebo versus Brivaracetam (BRV) 150 mg/day, the primary endpoint will be tested for Placebo versus BRV 5 mg/day. In case of significance, the three UMRS related secondary endpoints will be tested for Placebo versus BRV 5 mg/day, provided the previous is significant at 5 %. Secondary endpoints are tested in the following order: * Functional Disability * Stimulus Sensitivity * Myoclonus Patient Questionnaire; Test type: Superiority or Other; p = 0.806, stratified Wilcoxon Test — Tested at the 5 % level - given the primary endpoint testing Placebo versus Brivaracetam (BRV) 5 mg/day is significant at the 5 % level (hierarchical testing procedure); Estimates and confidence intevals are obtained from Hodges-Lehmann (unstratified); Hodges-Lehmann-estimator of difference = 0.00, 95% CI 2-sided [-33.33 to 18.75] — Difference versus Placebo

3. Secondary Outcome: Percent Change From Baseline to the End of Treatment Period on the Stimulus Sensitivity Score (Unified Myoclonus Rating Scale (UMRS) Section 3)
Description: The range for Stimulus Sensitivity Score is 0 (best) to 17 (worst). Percent change from Baseline = 100 X ((Baseline UMRS3 - Treatment UMRS3) / Baseline UMRS3). Baseline is defined as the last non-missing value prior to or on Randomization Visit.
Time Frame: Baseline to End of Treatment Period (Week 14 or Early Discontinuation Visit)
Population: The number of subjects is equal to the number of subjects in the Intent-To-Treat (ITT) population having non-missing post-baseline results for the percent change from baseline on the stimulus sensitivity score (UMRS section 3). In case a subject drops out, the result at Early Discontinuation Visit (EDV) is used.
Measure: Median (Full Range); unit: Percent change
Arm/Group | Placebo | Brivaracetam 5 mg/Day | Brivaracetam 150 mg/Day
Number analyzed (Participants) | 18 | 20 | 18
Percent change | 0.00 [-300.0 to 100.0] | 43.44 [-300.0 to 100.0] | 0.00 [-300.0 to 100.0]
Statistical Analysis 1: Comparison: Placebo vs Brivaracetam 150 mg/Day; Test type: Superiority or Other; p = 0.549, stratified Willcoxon Test — Tested at the 5 % level - given the Functional Disability Score comparing Placebo versus Brivaracetam (BRV) 150 mg/day is significant at the 5 % level (hierarchical testing procedure); Estimates and confidence intervals are obtained from Hodges-Lehmann (unstratified); Hodges-Lehmann-estimator of difference = 0.00, 95% CI 2-sided [-25.00 to 100.00] — Difference versus Placebo
Statistical Analysis 2: Comparison: Placebo vs Brivaracetam 5 mg/Day; Test type: Superiority or Other; p = 0.654, stratified Wilcoxon Test — Tested at the 5 % level - given the Functional Disability Score comparing Placebo versus Brivaracetam (BRV) 5 mg/day is significant at the 5 % level (hierarchical testing procedure); Estimates and confidence intervals are obtained from Hodges-Lehmann (unstratified); Hodges-Lehmann-estimator of difference = 0.00, 95% CI 2-sided [-50.00 to 66.67] — Difference versus Placebo

4. Secondary Outcome: Percent Change From Baseline to the End of Treatment Period on the Myoclonus Patient Questionnaire (Unified Myoclonus Rating Scale (UMRS) Section 1)
Description: The range for Myoclonus Patient Questionnaire is 0 (best) to 44 (worst). Percent change from Baseline = 100 X ((Baseline UMRS1 - Treatment UMRS1) / Baseline UMRS1). Baseline is defined as the last non-missing value prior to or on Randomization Visit.
Time Frame: Baseline to End of Treatment Period (Week 14 or Early Discontinuation Visit)
Population: The number of subjects is equal to the number of subjects in the Intent-To-Treat (ITT) population having non-missing post-baseline results for the percent change from baseline on the Myoclonus Patient Questionnaire (UMRS section 1). In case a subject drops out, the result at Early Discontinuation Visit (EDV) is used.
Measure: Median (Full Range); unit: Percent change
Arm/Group | Placebo | Brivaracetam 5 mg/Day | Brivaracetam 150 mg/Day
Number analyzed (Participants) | 17 | 20 | 18
Percent change | -9.68 [-125.0 to 63.0] | 0.00 [-95.0 to 55.6] | 5.41 [-24.0 to 100.0]
Statistical Analysis 1: Comparison: Placebo vs Brivaracetam 150 mg/Day; Test type: Superiority or Other; p = 0.037, stratified Wilcoxon Test — [p-value comment as in outcome 3, analysis 1]; Estimates and confidence intervals are obtained from Hodges-Lehmann (unstratified); Hodges-Lehmann-estimator of difference = 14.29, 95% CI 2-sided [-1.76 to 39.39] — Difference versus Placebo
Statistical Analysis 2: Comparison: Placebo vs Brivaracetam 5 mg/Day; Test type: Superiority or Other; p = 0.111, stratified Wilcoxon Test — [p-value comment as in outcome 3, analysis 2]; Estimates and confidence intervals are obtained from Hodges-Lehmann (unstratified); Hodges-Lehmann-estimator of difference = 10.00, 95% CI 2-sided [-5.56 to 30.00] — Difference versus Placebo

5. Secondary Outcome: Global Evaluation Score (Investigator) at the End of Treatment Period
Description: The Global Evaluation Scale Score (Investigator) ranges from 1 (Marked worsening) to 7 (Marked improvement).
Time Frame: End of Treatment Period (Week 14 or Early Discontinuation Visit)
Population: The number of subjects is equal to the number of subjects in the Intent-To-Treat (ITT) population having non-missing post-baseline results for the Global Evaluation Score (I-GES). In case a subject drops out, the result at Early Discontinuation Visit (EDV) is used.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Brivaracetam 5 mg/Day | Brivaracetam 150 mg/Day
Number analyzed (Participants) | 18 | 20 | 18
percentage of participants
  Marked improvement | 0 | 10.0 | 11.1
  Moderate improvement | 11.1 | 0 | 11.1
  Slight improvement | 33.3 | 30.0 | 33.3
  No change | 50.0 | 50.0 | 33.3
  Slight worsening | 0 | 10.0 | 5.6
  Moderate worsening | 0 | 0 | 5.6
  Marked worsening | 5.6 | 0 | 0
Statistical Analysis 1: Comparison: Placebo vs Brivaracetam 5 mg/Day; Test type: Superiority or Other; p = 0.931, Stratified Wilcoxon test — The Global Evaluation Scale by Investigator (I-GES) was compared between placebo and each dose at 5 % significance level independently from the previous secondary endpoints
Statistical Analysis 2: Comparison: Placebo vs Brivaracetam 150 mg/Day; P-value for pairwise comparison of each Brivaracetam dose versus Placebo; Test type: Superiority or Other; p = 0.253, Stratified Wilcoxon test — [p-value comment as in outcome 5, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from Visit 1 (Week -2) until final Visit 10 (Week 18).
Description: The Intent-To-Treat (ITT) population consists of all randomized subjects who took at least one dose of study medication.
Arm/Group | Placebo | Brivaracetam 5 mg/Day | Brivaracetam 150 mg/Day
Serious Adverse Events (participants affected / at risk) | 2/18 | 3/20 | 2/18
Other Adverse Events (participants affected / at risk) | 13/18 | 13/20 | 15/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=18) | Brivaracetam 5 mg/Day (N=20) | Brivaracetam 150 mg/Day (N=18)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Grand mal convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Status epilepticus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Myoclonic epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Attention-seeking behavior (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=18) | Brivaracetam 5 mg/Day (N=20) | Brivaracetam 150 mg/Day (N=18)
Granulocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram QT corrected interval prolonged (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0)
Middle ear inflammation (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (3) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 1 (1) | 3 (6)
Oedema peripheral (General disorders) | 1 (2) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatomegaly (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 3 (4) | 1 (1) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1) | 1 (3)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 2 (3) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Joint sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Weight increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Myoclonus (Nervous system disorders) | 1 (2) | 4 (4) | 3 (4)
Somnolence (Nervous system disorders) | 2 (2) | 3 (3) | 4 (7)
Headache (Nervous system disorders) | 7 (8) | 3 (4) | 2 (2)
Balance disorder (Nervous system disorders) | 0 (0) | 1 (1) | 2 (4)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1)
Grand mal convulsion (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Hyporeflexia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Complex partial seizures (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Coordination abnormal (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0) | 1 (2)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (3)
Nystagmus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 3 (4) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Myoclonic epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Aggression (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Bradyphrenia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Disorientation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Memory impairment (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Enuresis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Genital pruritus female (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days